CLINICAL TRIAL: NCT04636580
Title: The Effect of Parents' Presence and Their Anxieties on Children's Dental Anxiety During Dental Procedures: Controlled Clinical Trial
Brief Title: Parental Affect in Dental Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Responsible Party: Principal Investigator, Tugba Yiğit, Principal Investigator, Uşak University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UsakU5
Record Dates: First submitted 2020-11-05; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Behavior; Dental Anxiety
Keywords: Behaviour; Dental anxiety; Parental presence
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anxious parent (Experimental): Parents were divided into two groups anxious and non-anxious.
  Interventions: Behavioral: parent accompanying the child during treatment
- non-anxious parent (Experimental): Parents were divided into two groups anxious and non-anxious.
  Interventions: Behavioral: parent accompanying the child during treatment

INTERVENTIONS:
Behavioral: parent accompanying the child during treatment — After the parents were divided into two groups, anxious and non-anxious, the groups were equally divided randomly and the parents accompanied their children during the treatment

SUMMARY:
Background: To evaluate the effect of the anxiety of a parent accompanying a child on the child's anxiety during treatment.

Methods: Parents of 160 patients (4-8 years old) were divided into two groups anxious and non-anxious. Each groups had separated two randomized subgroups that with/without parents accompanied their children. At the first visit, participating children were examined while the behavior of the child during the examination was evaluated by a single pediatric dentist according to their heart rates measured by a portable pulse oximeter and the data were recorded (objective data).Forty-two children with a score of 1 and 4 on the Frankel Scale were excluded. After the parents were divided into two groups, anxious and non-anxious, the groups were equally divided randomly and the parents accompanied their children during the treatment.

Patients were recalled after one week for the treatment visit. Both groups were evaluated using the basic behavior technique. Compomer fillings were performed on children with infiltration anesthesia. The children's heart rates were measured by a portable pulse oximeter during treatment. Finally, the children were asked to express how they felt about the treatment by pointing out one of the faces on the Wong-Baker Faces Scale (subjective data). The children also rated the experience on the Frankel scale administered by the same operator.

ELIGIBILITY:
Inclusion Criteria:

* mentally and physically healthy children with caries requiring anesthesia and no previous dental experience were selected for the study

Exclusion Criteria:

* children with a score of 1 and 4 on the Frankel Scale were excluded.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
change in anxiety during the treatment according to the accompaniment of the anxious parent of the child | An average of 6 months
  The child's anxiety during examination was evaluated with a pulse oximeter. The child's anxiety during examination was evaluated with a pulse oximeter.

CONTACTS AND LOCATIONS:
Overall Officials: Esra OZGOCMEN, Dr., Principal Investigator — Uşak University
Locations (1):
- Tuğba YIGIT, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No